CLINICAL TRIAL: NCT07132567
Title: Assessment of Safety and Efficacy of Poteligeo Inj. 20 mg (Mogamulizumab) Through Use-result Surveillance
Status: Recruiting | Type: Observational
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Poteligeo PMS
Record Dates: First submitted 2025-07-22; First posted 2025-08-20 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Mycosis Fungoides; Sezary Syndrome
Keywords: Poteligeo; mycosis fungoides; Sezary syndrome
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome | interventions — mogamulizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Poteligeo 20mg — Poteligeo 20mg
  Other Names: Mogamulizumab

SUMMARY:
The purpose of this surveillance is to assess the safety and efficacy of Poteligeo Inj. 20 mg (mogamulizumab) in routine clinical settings.

DETAILED DESCRIPTION:
This post-marketing surveillance (PMS) is designed as an all-case investigation in accordance with the Korean Ministry of Food and Drug Safety (MFDS) re-examination requirements. It targets adult patients with mycosis fungoides (MF) or Sézary syndrome (SS) who have received at least one prior systemic therapy and are treated with mogamulizumab (POTELIGEO® Injection 20 mg) under the approved indication in Korea.

Primary Objective: To assess the safety of mogamulizumab for patients treated under the approved indication in Korea.

Secondary Objective: To assess the effectiveness of mogamulizumab for patients treated under the approved indication in Korea.

Exploratory Objective: To perform additional subgroup and exploratory analyses of effectiveness, including evaluation in special populations such as elderly patients, patients with renal or hepatic impairment, and those with a history of hematopoietic stem cell transplantation, treated under the approved indication in Korea

ELIGIBILITY:
Inclusion Criteria:

1. Adults 19 years of age or older
2. Individuals who are confirmed to have received administration of the study drug for the purpose of "the treatment for adult patients with fungoidal granuloma or Sezary syndrome who have received one or more systemic therapies," or who are considered to require administration of the study drug in the investigator's opinion
3. Individuals who (or whose legally acceptable representatives) signed the Consent to Use of Personal Information of their own free will for participation in this use-result surveillance

Exclusion Criteria

1. Patients with hypersensitivity to any ingredients of this drug
2. Patients who intend to use this drug for non-approved indications
3. Patients who participated in a pre-market clinical trial of the study drug and received administration of the study drug

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A person who has Mycosis fungoides and sezary syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Safety (Special situation, adverse event, symptom, or disease occurring during treatment with Poteligeo) | From first administration of Poteligeo through 90 days after the last dose
  Number of participants who experience any adverse event or special situation during Poteligeo treatment and up to 90 days after the last dose, as recorded in CRFs based on medical examinations or spontaneous reports.

SECONDARY OUTCOMES:
Change from baseline to after 8th administration in Global Response Score (GRS) | Baseline (Day 1, prior to first dose) and Week 24 (after completion of 8th administration)
  Change in Global Response Score (GRS) from baseline (before first dose) to after the 8th administration, assessing skin, nodes, blood, and viscera. CR/PR = Effective; SD/PD/Relapse = Ineffective.

CONTACTS AND LOCATIONS:
Overall Officials: HaeMi Park, Study Director — Kyowa Kirin Korea Co., Ltd.
Locations (5):
- South Korea (5):
  - Kosin University Gospel Hospital, Busan, Busan Metropolitan City
  - Chung-Ang University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.